CLINICAL TRIAL: NCT01439191
Title: An Open-Label Randomized Phase II Study of Cipterbin® or Cipterbin® in Combination With Vinorelbine in Patients With HER2/Neu-overexpressed Metastatic Breast Cancer (MBC)
Brief Title: Study of Cipterbin®, Used Alone or With Vinorelbine in Patients With HER2/Neu-overexpressed Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai CP Guojian Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C302MBCⅡ
Record Dates: First submitted 2011-09-21; First posted 2011-09-23 (Estimated); Last update posted 2011-09-23 (Estimated); Status verified 2005-06

CONDITIONS: Metastatic Breast Cancer
Keywords: HER2-Overexpressed
MeSH Terms: conditions — Breast Neoplasms | interventions — Vinorelbine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- combination agent group (Experimental)
  Interventions: Drug: humanized anti-HER2 antibody; Drug: Vinorelbine
- single agent group (Experimental): In this arm, patients would be treated with Cipterbin® for 12 or 24 weeks
  Interventions: Drug: humanized anti-HER2 antibody

INTERVENTIONS:
Drug: humanized anti-HER2 antibody — Initial dose of 4 mg/kg as an intravenous infusion over 90 minutes then at 2 mg/kg as an intravenous infusion over 30 minutes weekly for 12 weeks. For single agent group, patients with complete response, partial response or stable disease could be treated for 24 weeks.
  Other Names: brand name:Cipterbin®
Drug: Vinorelbine — Vinorelbine was administered weekly at a dose of 25 mg/m2 on day 1, 8 and 21 every 4 weeks
  Other Names: brand name:NAVELBINE®
  Arms: combination agent group

SUMMARY:
The HER2 gene (also known as HER2/neu and ErbB2 gene) is overexpressed in 20-30% of human breast cancers and leads to a particularly aggressive form of the disease. Trastuzumab,a humanized anti-HER2/neu receptor monoclonal antibody, has been proved a valuable treatment for HER2-positive breast cancer patients.The combination of trastuzumab with chemotherapy has been shown to increase both survival and response rate, in comparison to trastuzumab alone. CMAB302, a biosimilar of trastuzumab, was developed by Shanghai CP Guojian Pharmaceutical Co.Ltd. Efficacy and safety of CMAB302 as a single agent or in combination with vinorelbine were evaluated in patients with HER2-overexpressing metastatic breast cancer.

DETAILED DESCRIPTION:
The HER2 gene (also known as HER2/neu and ErbB2 gene) is overexpressed in 20-30% of human breast cancers and leads to a particularly aggressive form of the disease. Trastuzumab,a humanized anti-HER2/neu receptor monoclonal antibody, has been proved valuable treatment for HER2-positive breast cancer patients.The combination of trastuzumab with chemotherapy has been shown to increase both survival and response rate, in comparison to trastuzumab alone. CMAB302, a biosimilar of trastuzumab, was developed by Shanghai CP Guojian Pharmaceutical Co.Ltd. Previous Phase I study showed that CMAB302 was well tolerated as monotherapy and the pharmacokinetic data exhibited a non-linear profile over the dose range of 100 to 500 mg, similar to that of trastuzumab. In this study, efficacy and safety of CMAB302 as a single agent or in combination with vinorelbine were evaluated in patients with HER2-overexpressing metastatic breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* pathologic diagnosis breast cancer
* HER2+ status defined as IHC3+ Staining or in situ hybridization positive at least 1 measurable lesion as per RECIST criteria
* Adequate bone marrow function (absolute neutrophil count >1500/mm3, platelet count >100.000/mm3, hemoglobin >10gr/mm3)
* Adequate liver (bilirubin <1.0 times upper limit of normal and SGOT/SGPT <2.5 times upper limit of normal) and renal function (creatinine <1.5mg/dl)
* Adequate cardiac function (LVEF>50%). Normal electrocardiogram and absence of significant heart disease
* age from 18 to 70y
* Karnofsky performance score ≥ 60
* Life expectancy of greater than 3 months
* Negative HCG pregnancy test for premenopausal women of reproductive capacity and for women less than 12 months after the menopause.
* signed ICF

Exclusion Criteria:

* prior exposure vinorelbine for breast cancer
* prior exposure trastuzumab for breast cancer
* Prior chemotherapy and radiation therapy within the last 4 weeks before enrollment
* use of any other investigational agents within the last 4 weeks before enrollment
* symptomatic, central nervous system metastases
* Hypersensitivity to trial medications
* breastfeeding or pregnant

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2005-07; Primary Completion 2007-02 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Overall response rate | up to 24 weeks
  according to RECIST 1.0 (Response Evaluation Criteria In Solid Tumors)

SECONDARY OUTCOMES:
One-year survival rate | 1 year
Number of participants with adverse events | up to 24 weeks
  Adverse events was recorded according to NCI CTC 2.0 (National Cancer Institute common toxicity criteria).
Overall control of disease | up to 24 weeks
  defined as overall response rate plus stable disease, by RECIST 1.0

CONTACTS AND LOCATIONS:
Overall Officials: Yan Sun, PhD, Study Chair — Cancer Institute and Hospital, Chinese Academy of Medical Sciences; Yuankai Shi, PhD, Study Director — Cancer Institute and Hospital, Chinese Academy of Medical Sciences; Zefei Jiang, PhD, Principal Investigator — Hospital Affiliated to Academy Military Medical Science; Jun Ren, PhD, Principal Investigator — Peking University Cancer Hospital & Institute; Xichun Hu, PhD, Principal Investigator — Fudan University; Kai Li, PhD, Principal Investigator — Tianjin Medical University Cancer Institute and Hospital; Dong Wang, PhD, Principal Investigator — Daping Hospital & Research Institute of Surgery of the Third Military Medical University
Locations (1):
- Cancer Institute and Hospital, Chinese Academy of Medical Sciences, Beijing, China